CLINICAL TRIAL: NCT02065960
Title: Feasibility Study of the Role of Stereotactic Body Radiotherapy for the Treatment of Early Stage Breast Cancer
Brief Title: Feasibility Study of Stereotactic Body Radiotherapy for Early Breast Cancer
Acronym: ARTEMIS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juravinski Cancer Center (Other)
Collaborators: Juravinski Cancer Centre Foundation (Other); Canadian Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Julie Arsenault, MD, FRCPC, Clinical Research Fellow, Radiation Oncology, Juravinski Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-699
Record Dates: First submitted 2014-02-12; First posted 2014-02-19 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Breast Neoplasm
Keywords: Feasibility study; Early breast cancer; Stereotactic body radiotherapy; Cyberknife; Pre-operative radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic body radiotherapy (SBRT) (Experimental): Radiotherapy with SBRT to a dose of 40 Gy in 5 fractions delivered every other day over a period of 10-12 days, followed by breast conserving surgery.
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT)
  Other Names: Cyberknife

SUMMARY:
Most women with early breast cancer are treated with breast conserving therapy (BCT), consisting of breast conserving surgery (surgery to remove the cancer itself) followed by radiation to the breast. This treatment can take time and is associated with its own side effect profile. An innovative radiation technique called stereotactic body radiotherapy (SBRT) can deliver large doses of radiation precisely to the tumour while avoiding critical organs, therefore destroying the cancer and avoiding surgery altogether. SBRT has been successfully used for a number of cancers and it is proposed that it could be used to eradicate breast cancer. This feasibility study will investigate the feasibility and safety of treatment using SBRT in women with early stage breast cancer.

Thirty-two women age 70 years or older with early breast cancer will be treated with SBRT (5 treatments) followed by breast conserving surgery and hormonal therapy. An MRI and breast conserving surgery will be performed at 8-12 weeks after radiation to assess response to treatment. The primary outcome of the study will be feasibility, meaning the ability to deliver radiation treatment as planned. Secondary outcomes will include treatment related toxicity and pathological response.

If this study shows that SBRT can be used to treat patients primarily, it will lead to further evaluation of SBRT for early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women age ≥ 70 years;
* New histological diagnosis of invasive carcinoma of the breast, grade I or II, estrogen and progesterone receptor (ER and PR) positive, HER2 negative on needle biopsy and limited to Stage I (T1 N0 M0) on clinical and radiological assessment with MRI of the breasts and axillary ultrasound;
* Candidate for breast conserving surgery;
* Signed study consent form completed prior to study entry.

Exclusion Criteria:

* Breast cancer with disease within 5 mm from skin or chest wall;
* Previous or concomitant invasive malignancies treated within 5 years of study entry;
* Serious non-malignant disease (cardiovascular, pulmonary, systemic lupus or scleroderma), which would preclude to definitive radiation therapy;
* Psychiatric disorders, which would preclude from obtaining informed consent
* Geographic inaccessibility for follow-up

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility | At time of radiation treatment delivery
  The primary outcome for this study will be successful delivery of SBRT as per protocol without a major deviation.

SECONDARY OUTCOMES:
Acute Radiation Toxicity | Within 3 months from radiation
Late Radiation Toxicity | 3 months or more after radiation
Pathological Response | At time of surgery (10-12 weeks post-radiation)
Ipsilateral Breast Tumour Recurrence | At 5 years post-registration
Disease Free Survival | At 5 years post-registration

CONTACTS AND LOCATIONS:
Overall Officials: Julie Arsenault, MD, FRCPC, Principal Investigator — Juravinski Cancer Centre; Do-Hoon Kim, BASc, MD, MSc, FRCPC, Principal Investigator — Juravinski Cancer Centre; Timothy Whelan, BSc, BM,BCh, MSc, FRCPC, Principal Investigator — Juravinski Cancer Centre
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada